CLINICAL TRIAL: NCT07195201
Title: Prospective Evaluation of Onlay Restorations Produced by Additive and Subtractive Manufacturing in Vital Posterior Teeth: A Split-Mouth
Brief Title: Clinical Evaluation of Additive and Subtractive Onlay Restorations
Acronym: CIP-ONLAY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Tugba Erturk Avunduk (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Ayse Tugba Erturk Avunduk, Associate Professor, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-ONLAY-2025-V01; 2025-157 (Registry Identifier: Turkish Medicines and Medical Devices Agency (TITCK))
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: CAD-CAM; Prospective Study; 3D Printing; Clinical Assessment
Keywords: onlay restorations; cad-cam; additive manufacturing; 3D printing; FDI criteria

STUDY DESIGN:
Intervention Model Description: "randomized, controlled, double-blind, split-mouth design"
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind clinical trial. Participants and outcome assessors are blinded to the allocation of onlay restorations fabricated by additive or subtractive manufacturing. The care provider performing the intervention cannot be blinded due to the nature of the manufacturing process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Additive Manufacturing (3D Printing) Onlay Restorations (Experimental): Onlay restorations will be fabricated using additive manufacturing technology (3D printing) with a biocompatible permanent resin (Bego VarseoSmile TriniQ). Restorations will be designed based on digital intraoral scans and placed in vital posterior teeth. Clinical evaluations will be performed at baseline (1 week), 6 months, 12 months, and 18 months according to FDI criteria.
  Interventions: Device: 3D Printed Onlay Restoration
- Subtractive Manufacturing (CAD/CAM Milling) Onlay Restorations (Active Comparator): Onlay restorations will be fabricated using subtractive manufacturing technology (CAD/CAM milling) with hybrid ceramic blocks (GC Cerasmart 270). Restorations will be designed based on digital intraoral scans and placed in vital posterior teeth. Clinical evaluations will be performed at (1 week), 6 months, 12 months, and 18 months according to FDI criteria.
  Interventions: Device: CAD/CAM Onlay Restoration

INTERVENTIONS:
Device: 3D Printed Onlay Restoration — Onlay restorations will be fabricated using a 3D printer and a biocompatible permanent resin (Bego VarseoSmile TriniQ). Digital intraoral scans will be used for design. Restorations will be placed in vital posterior teeth and evaluated at (1 week), 6 months, 12 months, and 18 months according to FDI criteria.
  Other Names: Additive Manufacturing; Bego VarseoSmile TriniQ
  Arms: Additive Manufacturing (3D Printing) Onlay Restorations
Device: CAD/CAM Onlay Restoration — Onlay restorations will be fabricated using a CAD/CAM milling unit and hybrid ceramic blocks (GC Cerasmart 270). Digital intraoral scans will be used for design. Restorations will be placed in vital posterior teeth and evaluated at (1 week), 6 months, 12 months, and 18 months according to FDI criteria.
  Arms: Subtractive Manufacturing (CAD/CAM Milling) Onlay Restorations

SUMMARY:
The goal of this clinical trial is to learn whether onlay restorations produced by additive manufacturing [three-dimensional (3D) printing] and subtractive manufacturing [Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) milling] perform equally well in vital posterior teeth. The main questions it aims to answer are:

* Do 3D printed onlay restorations show similar marginal adaptation and clinical performance compared to CAD/CAM milled onlays?
* Are there any differences in biological compatibility, surface properties, or postoperative sensitivity between the two techniques over time? Researchers will compare onlay restorations fabricated with 3D printing and CAD/CAM milling using a split-mouth study design.

Participants will:

* Receive one onlay restoration produced by 3D printing and another produced by CAD/CAM milling, placed on opposite sides of the mouth
* Have checkups at baseline (1st week), 6 months, 12 months, and 18 months after treatment
* Be evaluated using the Fédération Dentaire Internationale (FDI) criteria for marginal adaptation, surface quality, anatomical form, and biological compatibility

DETAILED DESCRIPTION:
This prospective, randomized, split-mouth clinical trial is designed to evaluate the clinical performance of onlay restorations fabricated by two different digital manufacturing techniques-additive manufacturing (3D printing) and subtractive manufacturing (CAD/CAM milling)-in vital posterior teeth.

Each participant will receive two onlay restorations: one produced by CAD/CAM milling using hybrid ceramic blocks (GC Cerasmart 270) and one produced by 3D printing with a biocompatible permanent resin (Bego VarseoSmile TriniQ). The restorations will be placed in contralateral posterior teeth, allowing direct intra-individual comparison under identical oral conditions. Randomization will determine which tooth receives which manufacturing method.

The primary outcome of the study is marginal adaptation, assessed according to the Fédération Dentaire Internationale (FDI) World Dental Federation criteria. Secondary outcomes include surface quality, anatomical form, functional stability, postoperative sensitivity, color match, and biological compatibility. Clinical evaluations will be performed at baseline (1 week) and at 6 months, 12 months, and 18 months.

To minimize bias, participants and clinical evaluators will remain blinded to the type of restoration applied. Calibration sessions will be conducted for all evaluators to ensure consistency and reliability of outcome assessment. An independent statistician, blinded to group allocation, will perform the statistical analyses.

A total of 29 participants are expected to be enrolled, based on power analysis using G*Power software, which indicated that this sample size provides 85% power with a 95% confidence level. Inclusion criteria consist of adults aged 18-84 with vital posterior teeth requiring onlay restorations, without systemic disease or active periodontal pathology. Teeth with pulp vitality confirmed by thermal or electrical testing and with moderate structural loss suitable for onlay restorations will be included. Exclusion criteria include teeth with previous endodontic treatment, advanced periodontal disease, or a history of full-coverage prosthetic restoration.

All procedures will follow standardized clinical protocols, including tooth preparation, digital intraoral scanning, design with CAD software, manufacturing with either milling or 3D printing, and adhesive cementation. Adverse events such as restoration failure, pulp complications, or allergic reactions to materials will be documented and reported according to regulatory requirements.

This study is expected to provide robust, long-term clinical evidence comparing the performance of additively and subtractively manufactured onlay restorations, addressing a current gap in the literature. The results will contribute to evidence-based clinical decision-making in digital restorative dentistry and support the development of guidelines for material and technique selection.

ELIGIBILITY:
Inclusion Criteria:

Participant-Level Criteria

* Adults aged 18-84 years
* No active periodontal disease (probing depth ≤ 3 mm, no clinical attachment loss)
* No parafunctional habits such as bruxism, clenching, or foreign object chewing
* Willingness to attend regular follow-up visits during the study period
* Adequate oral hygiene status
* No history of systemic disease or medically stable condition if present
* No history of similar restorative procedures involving the target teeth Tooth-Level Criteria
* Vital posterior teeth (premolars or molars) confirmed by thermal or electric pulp testing; teeth requiring endodontic treatment or with necrosis will be excluded
* Permanent posterior teeth located in functional occlusion (premolar or molar region)
* Teeth with moderate structural loss suitable for onlay restorations, including mesio-occlusal (MO), disto-occlusal (DO), or mesio-occluso-distal (MOD) cavities with partial crown loss but sufficient remaining tooth structure not requiring full coverage
* Periodontally healthy teeth with no mobility, no clinical attachment loss, and probing depth ≤ 3 mm
* Teeth that can be matched in contralateral quadrants to allow split-mouth design (structurally and clinically comparable teeth)
* Teeth free from cracks, fractures, or internal resorption; supporting tissues without structural defects that may compromise restoration success
* Teeth with clearly defined preparation margins located in enamel or sound dentin; subgingival margins extending deep into the sulcus will not be included
* Teeth without previous extensive prosthetic restorations (crowns, inlays/onlays, or implant-supported restorations)
* Opposing natural teeth in stable occlusal contact with the restored tooth

Exclusion Criteria:

* Teeth with pulp necrosis or a history of endodontic treatment (previous root canal therapy or non-vital teeth)
* Teeth with excessive tissue loss requiring full crown coverage and unsuitable for onlay restoration
* Teeth presenting with cracks, fractures, internal or external resorption, or structural defects compromising prognosis
* Advanced periodontal disease, including clinical attachment loss, furcation involvement, mobility, or probing depth > 3 mm
* Teeth with subgingival cavity margins extending deep into the gingival sulcus, increasing periodontal risk
* Teeth with a history of fixed prosthetic restorations (previous crowns, inlays/onlays, or bridge restorations)
* Teeth lacking proximal contacts due to adjacent tooth absence, leading to compromised contact stability and occlusal load distribution
* Teeth in regions with orthodontic appliances or fixed retainers that may interfere with restorative procedures or evaluation
* Opposing teeth absent or lacking stable occlusal contact with the restoration site
* Patients with systemic diseases contraindicate elective dental treatment (e.g., uncontrolled diabetes, immunocompromised status)
* Pregnant or breastfeeding women
* Patients unable or unwilling to attend scheduled follow-up visits [baseline (1 week), 6 months, 12 months, and 18 months]

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional Properties of Onlay Restorations | Baseline (1 week), 6 months, 12 months, and 18 months after restoration placement
  Functional performance of onlay restorations, including marginal adaptation, fracture and retention of the material, proximal contact point, anatomical form, occlusion, and wear, will be assessed using the Fédération Dentaire Internationale (FDI) criteria. Restorations will be scored as clinically excellent, clinically good, clinically sufficient/satisfactory, or clinically poor/unacceptable. The proportion of restorations receiving clinically acceptable scores (scores 1-3) will be recorded.

SECONDARY OUTCOMES:
Esthetic Properties of Onlay Restorations | Baseline (1 week), 6 months, 12 months, and 18 months
  Esthetic properties, including surface gloss and texture, marginal discoloration, and color match, will be assessed using FDI criteria. Restorations will be scored as clinically excellent, clinically good, clinically sufficient/satisfactory, or clinically poor/unacceptable. The proportion of restorations receiving clinically acceptable scores (scores 1-3) will be recorded.

OTHER OUTCOMES:
Biological Properties of Onlay Restorations | Baseline (1 week), 6 months, 12 months, and 18 months
  Biological properties, including secondary caries, hard tissue defects at restoration margins, postoperative sensitivity, and pulpal status, will be evaluated clinically and radiographically according to FDI criteria. Restorations will be scored as clinically excellent, clinically good, clinically sufficient/satisfactory, or clinically poor/unacceptable. The proportion of restorations receiving clinically acceptable scores (scores 1-3) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Faculty of Dentistry, Department of Restorative Dentistry, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated, anonymized study results will be disseminated through scientific publications and conference presentations.

REFERENCES:
- [Background] Revilla-Leon M, Alonso Perez-Barquero J, Barmak AB, Agustin-Panadero R, Fernandez-Estevan L, Gomez-Polo M. Accuracy of Intraoral Scanner Systems for Fabricating Inlay, Onlay, and Veneer Restorations: A Systematic Review and Meta-Analysis. J Esthet Restor Dent. 2025 Mar;37(3):727-755. doi: 10.1111/jerd.13361. Epub 2024 Dec 11. PMID 39663747
- [Background] Weick A. Issues in overturning a medical model of social work practice. Soc Work. 1983 Nov-Dec;28(6):467-71. doi: 10.1093/sw/28.6.467. No abstract available. PMID 10264483
- [Background] Coskun E, Aslan YU, Ozkan YK. Evaluation of two different CAD-CAM inlay-onlays in a split-mouth study: 2-year clinical follow-up. J Esthet Restor Dent. 2020 Mar;32(2):244-250. doi: 10.1111/jerd.12541. Epub 2019 Oct 23. PMID 31642587
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36504246/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31642587/